CLINICAL TRIAL: NCT05231850
Title: A Phase II Study of Tislelizumab as Adjuvant Therapy for Patients With High-risk Stage Ⅱ and Stage Ⅲ Colon Cancer and Deficient Mismatch Repair or Microsatellite Instability.
Brief Title: A Phase II Study of Tislelizumab as Adjuvant Therapy for Patients With Stage Ⅱ and Stage Ⅲ Colon Cancer and dMMR/MSI.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Feng Wang, Doctor, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Wfeng-001
Record Dates: First submitted 2022-02-07; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab (Experimental): Tislelizumab
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — All eligible patients receive received 200 mg Tislelizumab intravenously every 3 weeks until disease progression, unacceptable adverse events (AEs) or withdrawal of consent.

SUMMARY:
10%-15% of early-stage colon cancers harbour either deficient mismatch repair (dMMR), microsatellite instability high (MSI-H) is characterised by high tumour mutational burden and increased lymphocytic infiltrate. Metastatic dMMR colon cancers are highly sensitive to immune checkpoint inhibition.The MSI phenotype is associated with a better prognosis than MSS in stage II and III CRCs. However, there are conflicting data about the benefit of adjuvant chemotherapy in this group of patients.

We are conducting a single arm study phase II trial to determine if the anti-PD-1 antibody Tislelizumab improves disease-free survival (DFS) in patients with high risk stage II and stage III dMMR/MSI-H colon cancer.

DETAILED DESCRIPTION:
This study is a phase II, single arm study with main purpose to evaluate the safety, tolerability and efficacy of Tislelizumab as adjuvant therapy for patients with high-risk stage Ⅱ and stage Ⅲ colon cancer and deficient mismatch repair or microsatellite instability.

Tumour MMR status will be routinely tested locally as per NICE guidelines (either in the pre-operative biopsy or resection specimen). Subjects whose tumours are dMMR can sign the main study consent and undergo the study screening procedures.All eligible patients receive received 200 mg Tislelizumab intravenously every 3 weeks until disease progression, unacceptable adverse events (AEs) or withdrawal of consent. The maximum duration of the trial intervention period was 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥18 years
2. ECOG PS 0/1
3. Histologically proven, high-risk stage II (i.e., T3 or T4, N0, M0) and III (i.e., any T, N1 or N2, M0) adenocarcinoma of the colon (as defined by the presence of the inferior pole of the tumour above the peritoneal reflection - that is, at least 15 cm from the anal margin).
4. Fully surgically resected tumour with clear resection margins (i.e., >1 mm)
5. Locally confirmed defective mismatch repair (dMMR) tumour (as defined by the lack of staining on either the pre-operative biopsy samples or resection specimens of at least one of the following proteins: MLH1 (mutL homolog 1), MSH2 (mutS homologue 2), MSH6 (mutS homolog 6).
6. Patients with testing that did not show dMMR (loss of MMR protein) are not eligible to participate; patients whose tumors show MSI-H by polymerase chain reaction (PCR)-based assay are not eligible to participate unless they also have MMR testing by IHC and are found to have dMMR (i.e. loss of one or more MMR proteins).
7. Absence of metastases as shown by post-operative CT scan.
8. No prior medical therapy (chemotherapy, immunotherapy, biologic or targeted therapy) or radiation therapy for the current colon cancer except for one cycle of mFOLFOX6.
9. Absence of major post-operative complications or other clinical conditions that, in the opinion of the investigator, would contraindicate adjuvant chemotherapy 8. Adequate hematological function defined by absolute neutrophil count (ANC) ≥1.5 × 109/L, platelet count ≥100 × 109/L, and hemoglobin ≥9 g/dL (blood transfusion before recruitment is allowed)
10. Adequate hepatic function defined by a total bilirubin level ≤1.5 × the upper limit of normal (ULN) range and AST and ALT levels ≤2.5 × ULN 10. Adequate renal function defined by an estimated creatinine clearance ≥30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method) 11. Negative serum or urine pregnancy test at screening for women of childbearing potential 12. Fertile men and women must agree to take highly effective contraceptive precautions during, and for 6 months after the last dose of chemotherapy or for 1 month after the last dose of Tislelizumab

Exclusion Criteria:

1. Rectal tumours (as defined by the presence of the inferior pole of the tumour below the peritoneal reflection - that is, <15 cm from the anal margin).
2. Administration of neoadjuvant systemic chemotherapy or radiotherapy before surgical resection of colon cancer
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
4. Has a history of non-infectious pneumonitis that required steroids; currently active non-infectious pneumonitis; or evidence of interstitial lung disease.
5. Has an active infection requiring systemic therapy or history of uncontrolled infection.
6. Pregnancy or lactation
7. Known alcohol or drug abuse
8. Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥3 NCI-CTCAE v5.0), any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma)
9. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication
10. Known history of colitis, pneumonitis and pulmonary fibrosis (for example, inflammatory bowel disease, uncontrolled asthma), which, in the opinion of the Investigator, might impair the subject's tolerance of trial treatment.
11. Any psychiatric condition that would prohibit the understanding or rendering of informed consent
12. Vaccination within 4 weeks of the first dose of Avelumab and while on trial is prohibited except for administration of inactivated vaccines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Primary End point: Disease Free survival [ Time Frame: 3 years ] | 3 years
  Disease-free survival (DFS) at 3 years. DFS is measured from the date of randomisation to the date of first relapse (radiological or clinical) or death from any cause.

SECONDARY OUTCOMES:
Overall survival | 5 years
  the time from randomization to death, from any cause
Incidence of adverse events | Up to 30 days after last treatment
  Incidence of adverse events